CLINICAL TRIAL: NCT00129818
Title: A Study to Evaluate the Effect of Famciclovir in Reducing Herpes Virus Shedding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CFAM810A2404
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Genital Herpes
Keywords: Genital herpes; viral shedding; famciclovir; Symptomatic genital herpes; Asymptomatic genital herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Famciclovir

INTERVENTIONS:
Drug: Famciclovir

SUMMARY:
The study is designed to assess the efficacy and safety of famciclovir 250 mg twice a day (bid) suppressive treatment in men and women with herpes virus type 2 (HSV-2) infection, with and without a reported history of genital herpes and with or without herpes virus type 1 (HSV-1) seropositivity.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females at least 18 years of age with HSV-2 seropositive serology with or without history of clinically diagnosed recurrent genital herpes

Exclusion Criteria:

* Pregnancy
* History of renal dysfunction
* Use of immunosuppressive therapy, including steroids (other than topical or inhaled), or use of probenecid
* Hypersensitivity to famciclovir, valacyclovir or drugs with similar chemical structure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Group 1. Reduction of HSV DNA PCR positive days in HSV-2 seropositive patients with a history of clinical genital herpes lesions
Group 2. Reduction of HSV DNA PCR positive days in HSV-2 seropositive patients without a history of clinical genital herpes lesions

SECONDARY OUTCOMES:
reduction of HSV DNA PCR positive days without lesions in HSV-2 seropositive patients with and without a history of clinical genital herpes lesions
quantitative HSV DNA PCR, during the days with positive HSV-2 shedding.
time to the first recurrence of genital herpes and number of genital herpes recurrence episodes
oral HSV-1 and/or HSV-2 shedding in HSV-1 and HSV-2 seropositive patients
reduction of HSV DNA PCR positive days with lesions in HSV-2 seropositive patients with and without a history of clinical genital herpes lesions

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Orlando Clinical Research Center, Orlando, Florida
  - IU Center for Clinical STD Research, Indianapolis, Indiana
  - UNC Clinical Research - Raleigh, Raleigh, North Carolina
  - Lynne Health Science Institute, Oklahoma City, Oklahoma
  - Westover Heights Clinic, Portland, Oregon
  - University of Washington - Virology Research Clinic, Seattle, Washington